CLINICAL TRIAL: NCT07036562
Title: Time-restricted Eating and High-intensity Interval Training for Long-term Improvement in Metabolic Health
Brief Title: Time-restricted Eating and High-intensity Interval Training for Metabolic Health in Adults With Overweight/Obesity
Acronym: TREHIIT-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 911308
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity
Keywords: time-restricted eating; high-intensity interval training; exercise; diet; metabolic health; lifestyle intervention
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating and high-intensity interval training (Experimental): 12 months of periodised time-restricted eating and high-intensity interval training with digital follow-up
  Interventions: Behavioral: Time-restricted eating and high-intensity interval training
- Control (No Intervention): No intervention or follow-up. Habitual lifestyle

INTERVENTIONS:
Behavioral: Time-restricted eating and high-intensity interval training — 1-month intense periods of maximal daily eating window of 10 hours and high-intensity interval training (three weekly, unsupervised, aerobic exercise sessions performed at > 90 % heart rate maximum), separated by 3-month maintenance periods of time-restricted eating on 5 days per week and minimum 1 HIIT session per week. Each exercise session will last for 33-38 minutes. Participants will receive digital follow-up once weekly during intense periods, and once monthly during maintenance periods. The intervention period will be 12 months in total.
  Arms: Time-restricted eating and high-intensity interval training

SUMMARY:
This study will investigate the effects of 12 months periodised time-restricted eating combined with high-intensity interval training compared with a control group on fat mass in adults with overweight/obesity. Participants in the intervention group will complete the intervention remotely and will receive follow-up by telephone. Before randomisation, after 6 months and after 12 months, the investigators will measure the participants' body composition, physical fitness, fasting blood glucose and insulin, blood lipids, and blood pressure. Physical activity, diet, sleep quality, appetite, and adherence to the intervention will also be measured. Secondary sub-analyses of sex differences in the responses to the intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 27 kg/m²
* Able to walk or ride a bike > 60 min

Exclusion Criteria:

* On-going pregnancy
* Lactation within 24 weeks of study commencement
* High-intensity exercise ≥ 1/week
* Habitual eating window ≤12 hours/day
* Taking hypertension, glucose-, or lipid-lowering drugs
* Body mass variation ≥ 4 kg three months prior to study commencement
* Known diabetes mellitus (type 1 or 2) or cardiovascular disease
* Working night shifts

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Total fat mass | From baseline to after 12 months
  Change in total fat mass measured with bioelectrical impedance analysis

SECONDARY OUTCOMES:
Blood glucose | From baseline to after 6 months and after 12 months
  Fasting concentration of plasma glucose
Total fat mass | From baseline to after 6 months
  Change in total fat mass measured with bioelectrical impedance analysis
Insulin | From baseline to after 6 months and after 12 months
  Fasting concentration of plasma insulin C-peptide
Average glucose levels | From baseline to after 6 months and after 12 months
  Glycated haemoglobin (HbA1c)
Blood cholesterol | From baseline to after 6 months and after 12 months
  Total fasting cholesterol in blood
LDL-cholesterol | From baseline to after 6 months and after 12 months
  Fasting low-density lipoprotein-cholesterol in blood
HDL-cholesterol | From baseline to after 6 months and after 12 months
  Fasting high-density lipoprotein-cholesterol in blood
Triglycerides | From baseline to after 6 months and after 12 months
  Fasting triglycerides in blood
Cardiorespiratory fitness | From baseline to after 6 months and after 12 months
  Peak oxygen uptake at a maximum effort test, measured in mL/min/kg and L/min
Insulin sensitivity | From baseline to after 6 months and after 12 months
  Homeostatic model assessment for insulin resistance (HOMA-IR): 1.5 + fasting plasma glucose (mmol/L) x fasting plasma insulin C-peptide (pmol/L)/2800
Body mass | From baseline to after 6 months and after 12 months
  In kg, estimated with bioelectrical impedance analysis
Fat-free mass | From baseline to after 6 months and after 12 months
  In kg, estimated with bioelectrical impedance analysis
Visceral fat area | From baseline to after 6 months and after 12 months
  In cm2, estimated with bioelectrical impedance analysis
Systolic blood pressure | From baseline to after 6 months and after 12 months
  Average of three measurements during rest in seated position, in mmHg
Diastolic blood pressure | From baseline to after 6 months and after 12 months
  Average of three measurements during rest in seated position, in mmHg
Resting heart rate | From baseline to after 6 months and after 12 months
  Average of three measurements during rest in sitting position, in beats/min
Physical activity levels | From baseline to after 6 months and after 12 months
  International Physical Activity Questionnaire
Diet intake | During baseline week, after 4, 13, 30, and 50 weeks.
  3-day diet diaries (two weekdays and one weekend day) with online diet diary.
Sleep quality | From baseline to after 6 months and after 12 months
  The Pittsburgh Sleep Quality Index questionnaire

OTHER OUTCOMES:
Adherence to high-intensity interval training | 12 months
  Number of completed exercise sessions out of those prescribed, in percentage
Compliance to high-intensity interval training | 12 months
  Exercise intensity measured with pulse sensor. Heart rate percentage of individual heart rate maximum.
Adherence to time-restricted eating | During baseline week, after 4, 13, 30, and 50 weeks.
  Average number of days per week a daily eating window of 10 hours or less was achieved
Compliance to time-restricted eating | During baseline week, after 4, 13, 30, and 50 weeks.
  Average daily eating window, self-reported in hours/day
Perception of intervention and digital follow-up | After 12 months
  Qualitative interviews with selected participants to explore barriers and motivators
Sex differences | From baseline to after 6 months and after 12 months
  Sub-analyses of sex differences in the effectiveness of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of circulation and medical imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified individual participant data (IPD) collected in the study available to other researchers. We will upload a data set in an open access repository.
  We will only share IPD that cannot be used to identify individuals.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will become available at the time of publication of the results from the study.
Access Criteria: Open access